CLINICAL TRIAL: NCT05191420
Title: BECAUSE YOU MATTER: Conversations You Want About COVID-19
Brief Title: Conversations You Want About Corona Virus Disease (COVID-19)
Acronym: COVID-19
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00075790
Record Dates: First submitted 2022-01-11; First posted 2022-01-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Covid19
Keywords: Vaccines
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual topical discussion guide: Study will pilot test this virtual topical discussion guide to assess feasibility and acceptability by diverse patient populations.

SUMMARY:
Web-enabled virtual topical guide: develop virtual conversations for each concern and intensity level

DETAILED DESCRIPTION:
Study will pilot test the virtual topical discussion guide with diverse health care professions and community members to confirm it is clear, relevant, understandable, and culturally appropriate

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* English or Spanish speaking only

Exclusion Criteria:

* less than 18 years of age
* not English or Spanish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diverse health care professions and community members
Sampling Method: Probability Sample
Enrollment: 23000 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time spent with the guide | Week 4
  Time spent with the guide
Number of clinics viewed in the guide | Week 4
  Number of clinics viewed in the guide
Number of content areas accessed | Week 4
  Number of content areas accessed
Time spent with each content area | Week 4
  Time spent with each content area
Helpfulness of Tool | Week 4
  How helpful was this tool in your decision-making, ranging from 1 not at all helpful to 5 incredibly helpful
Number of Subjects saving responses | Week 4
  Individuals will have the ability to send their guide responses to themselves for later use

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Poehling, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No